CLINICAL TRIAL: NCT04939363
Title: A Prospective, Phase-II Study to Evaluate the Efficacy and Safety of Obinutuzumab, Ibrutinib, and Venetoclax in Patients With Richter's Syndrome. GIVeRS Protocol: On Behalf of the Israeli CLL Study Group
Brief Title: A Study to Evaluate Efficacy & Safety of Obinutuzumab, Ibrutinib, and Venetoclax in Richter's Syndrome;
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA-002804
Record Dates: First submitted 2021-06-06; First posted 2021-06-25 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-11

CONDITIONS: Richter's Syndrome
MeSH Terms: interventions — obinutuzumab; ibrutinib; venetoclax

STUDY DESIGN:
Intervention Model Description: non-randomized, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination of Ibrutinib, Venetoclax and Obinutuzumab (Experimental): 1. Obinutuzumab intravenous infusion:
     Cycles 1: Day 1: Obinutuzumab 100 mg Day 1 (or 2): Obinutuzumab 900 mg Day 8: Obinutuzumab 1000 mg Day 15: Obinutuzumab 1000 mg Cycles 2-6: Day 1: Obinutuzumab 1000 mg The first infusion of Obinutuzumab may be administered at the full dose (1000 mg) on day 1 of cycle 1, if the infusion of a test-dosage of 100 mg is well tolerated by the patient. Alternatively, if the first 100 mg infusion on day 1 is not well tolerated, the remaining 900 mg of the first dose should be administered on day 2.
  2. Ibrutinib PO 560mg daily starting on cycle 1 day 1 for 12 cycles.
  3. Venetoclax with an accelerated ramp-up and close inpatient TLS monitoring starts on cycle 1 day 15 to the target dose of 400mg daily for a total of 12 cycles:
  Cycle 1: Day 15: Venetoclax 20 mg Days 16-17: Venetoclax 50 mg Days 18-21: Venetoclax 100 mg Days: 22-28: Venetoclax 200 mg Cycles 2-12: Days 1-28: Venetoclax 400 mg
  Interventions: Combination Product: Obinutuzumab with Ibrutinib and Venetoclax

INTERVENTIONS:
Combination Product: Obinutuzumab with Ibrutinib and Venetoclax — 1. Obinutuzumab intravenous infusion:
  2. Ibrutinib PO 560mg daily starting on cycle 1 day 1 for 12 cycles.
  3. Venetoclax with an accelerated ramp-up and close inpatient Tumor Lysis Syndromes (TLS) monitoring starts on cycle 1 day 15 to the target dose of 400mg daily for a total of 12 cycles:

SUMMARY:
Richter's syndrome (RS) is a life-threatening complication of chronic lymphocytic leukemia (CLL). It is associated with a switch in histopathology and biology, generally with a transformation of the original CLL clone to diffuse large B-cell lymphoma (DLBCL). The development of RS is accompanied by the onset of B symptoms, rapid growth of lymphadenopathy, extra-nodal disease, significant elevations of lactate dehydrogenase (LDH), and associated multi-organ dysfunction from invasive or obstructive processes RS occurs in 2-10% of CLL patients with an incidence rate of 0.5% per year. The molecular pathogenesis of RS involves inactivation of the tumor protein p53 (TP53) tumor suppressor gene in 50-60% of cases and activating aberrations of NOTCH1 and myelocytomatosis oncogene (MYC) in about 30% of cases. .

These distinct molecular footprints of RS are chemoresistance leading to an aggressive clinical course with low response rates and poor outcomes.Taking into consideration that in addition to the underlying aggressive disease, most RS patients are often at an advanced age and suffer from numerous other comorbidities. Additionally, intensive chemotherapy regimens are highly toxic to this population group and lead to excessive treatment-related morbidity. Enrolling DLBCL-RS patients in clinical trials is therefore justifiable, particularly those with RS that is clonally related to the predisposed underlining CLL disease. Due to the poor activity of immunochemotherapy, the possibility of using novel agents in the treatment of RS is of great interest.

The toxicity and the efficacy of the combination of cluster of anti differentiation antigen 20 (anti-CD20) antibody (e.g. Obinutuzumab or Rituximab) with Ibrutinib and/or Venetoclax have been already reported in both relapsed and naïve patients with CLL. The use of these three agents in combination is highly active in CLL and has manageable side effects. In addition, recent reports showed that treatment with Ibrutinib or Venetoclax as a single drug are active in RS.

Herein the investigators propose a phase 2, open-label, non-randomized, single arm, multi-center study aiming to assess the safety and efficacy with the combination of Ibrutinib, Venetoclax and Obinutuzumab in patients with RS

.

DETAILED DESCRIPTION:
Richter's syndrome (RS) is a life-threatening complication of chronic lymphocytic leukemia (CLL). It is associated with a switch in histopathology and biology, generally with a transformation of the original CLL clone to diffuse large B-cell lymphoma (DLBCL). The development of RS is accompanied by the onset of B symptoms, rapid growth of lymphadenopathy, extra-nodal disease, significant elevations of LDH, and associated multi-organ dysfunction from invasive or obstructive processes.

Previous research has increased general knowledge on the distinct evolutionary patterns of RS and provided a deeper understanding of the risk factors and molecular events predisposing to transformation. However, currently there're main few targetable aberrations and treatment is largely ineffective with a dismal prognosis leaving these patients with a high unmet medical need for better treatment strategies.

RS occurs in 2-10% of CLL patients with an incidence rate of 0.5% per year. The molecular pathogenesis of RS involves inactivation of the TP53 tumor suppressor gene in 50-60% of cases and activating aberrations of NOTCH1 and MYC in about 30% of cases.

These distinct molecular footprints of RS are chemoresistance leading to an aggressive clinical course with low response rates and poor outcomes. Patients with RS are usually excluded from clinical trials and there is no established standard of care in the treatment of RS today.

A number of chemotherapy regimens have been evaluated in the treatment of DLBCL-RS resulting in overall responses ranging between 40%-60% which are short lived with disappointing Progression Free Survival (PFS) and Overall Survival (OS) ranging between 3 - 10 and 6 - 21 months, respectively.

In Israel the current treatment strategy used for newly diagnosed DLBCL-RS is an anthracycline-based regimen, rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP). This treatment regimen has shown poor efficacy in a cohort study of 15 DLBCL-RS patients prospectively evaluated by a German CLL study group trial. The ORR was 67% with only 7% Complete Response (CR). The median PFS and median OS were 10 and 21 months, respectively in these patients. In terms of the safety profile of R-CHOP for patients with DLBCL-RS or CLL patients, 15 of the 60 (25%) patients enrolled in this study had therapy discontinued earlier than planned because of the treatment-related toxicity.

Taking into consideration that in addition to the underlying aggressive disease, most RS patients are often at an advanced age and suffer from numerous other comorbidities, therefore only 10%-15% of patient scan undergo the potentially curative allogeneic Hematopoietic Stem Cell Transplantation (HSCT). Additionally, intensive chemotherapy regimens are highly toxic to this population group and lead to excessive treatment-related morbidity. Enrolling DLBCL-RS patients in clinical trials is therefore justifiable, particularly those with RS that is clonally related to the predisposed underlining CLL disease. Due to the poor activity of immunochemotherapy, the possibility of using novel agents in the treatment of RS is of great interest.

The toxicity and the efficacy of the combination of anti-CD20 antibody (e.g. Obinutuzumab or Rituximab) with Ibrutinib and/or Venetoclax have been already reported in both relapsed and naïve patients with CLL. The use of these three agents in combination is highly active in CLL and has manageable side effects. In addition, recent reports showed that treatment with Ibrutinib or Venetoclax as a single drug are active in RS.

Herein the investigators propose a phase 2, open-label, non-randomized, single arm, multi-center study aiming to assess the safety and efficacy with the combination of Ibrutinib, Venetoclax and Obinutuzumab in patients with RS.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years of age or older.
2. Patients with histopathological confirmation of Richter's transformation into diffuse large B-cell lymphoma (DLBCL).
3. Subjects must have at least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma. The site of disease must be greater than 1.5 cm in the long axis regardless of short axis measurement or greater than 1.0 cm in the short axis regardless of long axis measurement, and clearly measurable in 2 perpendicular dimensions.
4. Eastern Cooperative Oncology Group (ECOG) status 0 to 2; ECOG 3 is only permitted if related to RS.
5. Adequate renal function, as indicated by an estimated creatinine clearance higher than 30 ml/min, adequate platelet count > 25 x 109/L, adequate liver function as indicated by total bilirubin < x 2 and Alanine transaminase (ALT) < x 2.5 of the institutional upper normal levels, unless directly attributable to the RS or to Gilbert's Syndrome.
6. Negative serological testing for hepatitis B (anti-hepatitis Bc negative, patients positive for anti-hepatitis Bc may be included if Polymerase chain reaction (PCR) for HBV DNA is negative) and negative HIV test performed within 6 weeks prior to enrollment.
7. Ability and agreement to provide written informed consent and to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Diagnosed or treated for malignancy other than DLBCL-RS or CLL/Small Lymphocytic Lymphoma (SLL) , except:

   1. Malignancy treated with curative intent and with no known active disease present at enrollment.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna melanoma without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease.
2. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of enrollment, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
3. Requires anticoagulation with coumadin or equivalent vitamin K antagonists (e.g., phenprocoumon).
4. Requirement of therapy with strong CYP3A4 and CYP3A5 inhibitors/inducers.
5. Documented resistance to Ibrutinib and/or Venetoclax.
6. Pregnant women and nursing mothers (a negative pregnancy test is required for all women of childbearing potential within 7 days before start of treatment; further pregnancy testing will be performed regularly).
7. Fertile men or women of childbearing potential unless:

   1. surgically sterile or ≥ 2 years after the onset of menopause
   2. Willing to use two methods of reliable contraception including one highly effective contraceptive method (Pearl Index <1) and one additional effective (barrier) method during study treatment and for 18 months after the end of study treatment.
8. Positive serological test for human immunodeficiency virus (HIV) or active Hepatitis C Virus (HCV; RNA polymerase chain reaction [PCR]-positive) or active Hepatitis B Virus (HBV; DNA PCR-positive) infection or any uncontrolled active systemic infection. Subjects with PCR-negative HBV and HCV are permitted in the study.
9. Legal incapacity.
10. Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of Ibrutinib capsules, or put the study outcomes at undue risk.
11. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment parameters-Safety | Up to 3 years from last patient enrollment
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment parameters.
Overall Response Rate -ORR | Up to 6 months from last patient enrollment
  Overall Response Rate (ORR) defined as the sum of partial response (PR) and complete response -(CR) determined by PET-CT imaging at 6 months according to the 2014 Lugano criteria assessing FluoroDeoxyGlucose (FDG)-Positron emission tomography-computed tomography (PET/CT) in lymphoma

SECONDARY OUTCOMES:
Progression-free survival -PFS | Up to 3 years from last patient enrollment
  Progression-free survival (PFS) defined as the time from the date of treatment initiation to the date of progression according to the Lugano criteria
Overall survival -OS | Up to 3 years from last patient enrollment
  Overall survival (OS) defined as the time from treatment initiation to death from any cause. If the subject is alive or the vital status is unknown, then the subject will be censored at the date the subject was last known to be alive.
Incidence of adverse events | Up to 3 years from last patient enrollment
  Incidence of adverse events, defined as the occurrence of all grades of toxicity (using CTCAE version 5.0) with special emphasis on adverse events of special interest (AESI) and their relationship to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Herishanu, Prof, Principal Investigator — TASMC; Tamar Tadmor, Prof, Principal Investigator — Bnai Zion Medical Center; Ohad Benjamini, Dr., Principal Investigator — Sheba Medical Center; Neta Goldschmidt, Prof, Principal Investigator — Hadassah Medical Organization
Locations (4):
- Israel (4):
  - Bnai Zion Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - TASMC, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No